CLINICAL TRIAL: NCT01706276
Title: MASIMO Radical 7 and Laboratory Measurement
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Other Study IDs: TJMZK20120902
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Major Hepatic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Present study aimed to evaluate the accuracy of Masimo Radical 7 to monitor hemoglobin concentrations through compared with laboratory measurement during major hepatic surgery, and to determine the source of discordance between two methods.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* American Society of Anesthesiologists Physical Status Ⅰor Ⅱ
* scheduled for potentially hemorrhagic major hepatic resection under general anesthesia
* requiring an arterial line

Exclusion Criteria:

* coagulopathy
* hemoglobinopathy
* cardiac dysrhythmias
* arrhythmia
* intracardiac shunt
* heart valve diseases
* tinea unguium
* arterio puncture failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, American Society of Anesthesiologists Physical Status Ⅰor Ⅱ, scheduled for potentially hemorrhagic major hepatic resection under general anesthesia and requiring an arterial line
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin measurement using the Masimo device | 0.5h after skin incision

SECONDARY OUTCOMES:
Change of Hemoglobin measurement using the Masimo device | 1h and 3h after skin incision

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China